CLINICAL TRIAL: NCT04505670
Title: The Effect of Donepezil on Wound Healing
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Stephen Wills, Principal Investigator, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SH2019-8
Record Dates: First submitted 2020-03-05; First posted 2020-08-10 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Wound Heal
MeSH Terms: interventions — Donepezil; Zinc Oxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Donepezil and Topical Zinc Oxide (Experimental): donepezil 5mg daily and topical zinc oxide 20% three times daily
  Interventions: Drug: Donepezil; Drug: Topical Zinc Oxide
- Placebo and Topical Zinc Oxide (Placebo Comparator): Placebo daily and topical zinc oxide 20% three times daily
  Interventions: Drug: Placebo oral tablet; Drug: Topical Zinc Oxide

INTERVENTIONS:
Drug: Donepezil — donepezil orally 5mg
  Arms: Donepezil and Topical Zinc Oxide
Drug: Placebo oral tablet — Placebo
  Arms: Placebo and Topical Zinc Oxide
Drug: Topical Zinc Oxide — Topical Zinc Oxide 20%

SUMMARY:
The purpose of the study is to test effectiveness of donepezil to improve wound healing in patients with diabetic wounds that have not healed with standard treatment.

DETAILED DESCRIPTION:
The study will be a randomized double blind study whereby patients with refractory diabetic wound healing over 3-6 months will be randomized to ascertain the effect of donepezil (administration of 5 mg to 10 mg of donepezil daily, orally, over 6 week period) on clinical wound healing reflecting correction of diabetic microvascular disease of non-healing wounds. The subjects will be recruited from the University of Maryland Shore Medical Center at Easton's emergency room and inpatients. Subjects will also be recruited from University of Maryland Shore Medical Group Wound Care and University of Maryland Baltimore Washington Medical Center's Vascular Clinic.

20 patients with Type 2 Diabetes Mellitus (Adult Onset Diabetes Mellitus) and non-healing ulcers/ wounds refractory to management with topical preparation and local debridement over a 3 to 6 month period prior will randomized to treatment or control group. The study group will be treated with oral donepezil (5 to 10 mg ). After 3 days of treatment, the dose of donepezil or placebo will be increased to 10 if no improvements are noted in skin integrity in the feet or lower extremity. Improvements in capillary refill and vascular edema will determine increase of donepezil from 5 to 10 mg. All patients will receive topical zinc oxide 20% topically three times a day, an effective topical management of diabetic wounds. Measurement of wound size and depth will be made prior to treatment. Additionally a color photograph will be obtained to compare with wound appearance in 6 weeks.

As many patients as required to meet the enrollment numbers shall be screened. Patients will be monitored daily for blood pressure, glucose levels and heart rate, during the period of hospitalization. Adjustments in insulin or oral hypoglycemic, blood pressure and heart rate control medications will occur during this time. Follow up visits will be made as required and at the end of week 6.

Donepezil shall be orally administered to the study group. Control group will get an orally administered placebo which is an inert compound, lactulose.

Wk0 will be the randomization visit. The patients will take the drug for 6 weeks and the last follow up visit will be the last day of week 6. Follow up at 6 weeks will occur at Shore Rehab at Easton.

Any anticholinergic drugs will be eliminated from the patients' medical regimen with the exception for inhaled anticholinergic. There is no known major contraindication of acetylcholinesterase inhibitors (like for eg: galantamine, rivastigmine and donepezil) Patients shall be monitored closely for vagotonic effect. Acetylcholine is known to have a vagotonic effect lowering heart rate and blood pressure. Therefore, during the course of administration of the drug close attention to heart rate and blood pressure will be a significant part off the clinical management of patients. If the patients are on beta blockers, their beta blocker dose will be closely monitored and adjusted as required.

H2 antagonist will be used to guard against any possible GI bleed, Pepcid 20mg a day.

Patient will be observed for seizures. The patients will be examined for pulmonary exacerbation during treatment in the hospital. If the pulmonary status deteriorates they will be eliminated from the study. The medication administration will not start sooner than 24 hrs after surgery. Patients shall be observed for exaggerated response from anesthesia.

Photographs of the diabetic wound/ ulcer and HgbA1C will be obtained on introduction to study and obtained at completion at 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 20
* diagnosed with Diabetes Mellitus

Exclusion Criteria:

* under the age of 20
* pregnant of lactating
* lactose intolerance
* allergy to donepezil
* prothrombin time and international normalized ratio value greater than 1.25
* Pre Menopausal women/ Women of childbearing potential

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-08-30 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in depth wound | 2-4 weeks
  Wound will be measured in centimeters and assessed for change.
Change in diameter of the wound | 2-4 weeks
  Wound will be measured in centimeters and assessed for change.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Shore Medical Center at Easton, Easton, Maryland, United States

IPD SHARING:
Plan to Share IPD: No